CLINICAL TRIAL: NCT00069784
Title: A Multicenter, International Randomized, 2x2 Factorial Design Study to Evaluate the Effects of Lantus (Insulin Glargine) Versus Standard Care, and of Omega-3 Fatty Acids Versus Placebo, in Reducing Cardiovascular Morbidity and Mortality in High Risk People With Impaired Fasting Glucose (IFG), Impaired Glucose Tolerance (IGT) or Early Type 2 Diabetes Mellitus: The ORIGIN Trial (Outcome Reduction With Initial Glargine Intervention)
Brief Title: The ORIGIN Trial (Outcome Reduction With Initial Glargine Intervention)
Acronym: ORIGIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: LTS6035; HOE901/4032 (Other: previous Aventis study number)
Record Dates: First submitted 2003-10-01; First posted 2003-10-06 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Impaired Fasting Glucose (IFG); Impaired Glucose Tolerance (IGT)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance | interventions — Insulin Glargine; Docosahexaenoic Acids; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Insulin glargine + omega-3 polyunsaturated fatty acids (Experimental): * Insulin glargine once daily by subcutaneous injection in a titrated regimen targeting a fasting plasma glucose (FPG) level of ≤95 mg/dL (5.3 mmol/L)
  * One capsule of omega-3 polyunsaturated fatty acids once daily
  Interventions: Drug: insulin glargine (HOE901); Drug: omega-3 polyunsaturated fatty acids (PUFA); Device: reusable pen device for insulin injection
- Insulin glargine + placebo (Experimental): * Insulin glargine once daily by subcutaneous injection in a titrated regimen targeting a fasting plasma glucose (FPG) level of ≤95 mg/dL (5.3 mmol/L)
  * One capsule of placebo once daily
  Interventions: Drug: insulin glargine (HOE901); Drug: placebo; Device: reusable pen device for insulin injection
- Standard care + omega-3 polyunsaturated fatty acids (Experimental): • One capsule of omega-3 polyunsaturated fatty acids once daily
  Interventions: Drug: omega-3 polyunsaturated fatty acids (PUFA)
- Standard care + placebo (Placebo Comparator): • One capsule of placebo once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: insulin glargine (HOE901) — Cartridges for use in a pen device, each containing 3 mL of insulin glargine 100 U/mL solution for injection
  Other Names: Lantus®
  Arms: Insulin glargine + omega-3 polyunsaturated fatty acids; Insulin glargine + placebo
Drug: omega-3 polyunsaturated fatty acids (PUFA) — Gelatin capsules (containing icosapent ethyl esters 465 mg and doconexent ethyl esters 375 mg) for oral administration
  Other Names: Omacor®
  Arms: Insulin glargine + omega-3 polyunsaturated fatty acids; Standard care + omega-3 polyunsaturated fatty acids
Drug: placebo — Matching placebo gelatin capsules (containing olive oil) for oral administration
  Arms: Insulin glargine + placebo; Standard care + placebo
Device: reusable pen device for insulin injection
  Other Names: OptiPen® Pro 1
  Arms: Insulin glargine + omega-3 polyunsaturated fatty acids; Insulin glargine + placebo

SUMMARY:
The primary objectives of the ORIGIN study were:

* To determine whether insulin glargine-mediated normoglycemia can reduce cardiovascular morbidity and/or mortality in people at high risk for vascular disease with either Impaired Fasting Glucose (IFG), Impaired Glucose Tolerance (IGT) or early type 2 diabetes;
* To determine whether omega-3 fatty acids can reduce cardiovascular mortality in people with IFG, IGT or early type 2 diabetes.

The secondary objectives of the insulin glargine study were to determine if insulin glargine-mediated normoglycemia can reduce:

* total mortality (all causes);
* the risk of diabetic microvascular outcomes;
* the rate of progression of IGT or IFG to type 2 diabetes.

DETAILED DESCRIPTION:
The ORIGIN study was conducted by the Population Health Research Institute in Hamilton, Ontario (Canada), working in conjunction with the sponsor, and an independent Steering Committee.

Routine visits were to occur at 2, 4, 8, and 16 weeks following randomization, then every four months for the rest of the study, for all participants

The duration of the study was based on the number of events observed (event-driven study) and was originally planned to be 5 years. In 2008-2009 ORIGIN's follow-up was extended by approximately 2 years, because of published literature of completed studies suggesting that a longer period of effective glycemic contrast between treatments might be needed to see an effect on cardiovascular events.

ELIGIBILITY:
Inclusion criteria:

I1. Individuals with IFG and/or IGT, or early diabetes, as defined below.

Glucose tolerance status was determined by a 75 g oral glucose tolerance test (OGTT) that was performed fasting (ie, no consumption of food or beverage other than water for at least 8 hours) at the time of screening for all candidates who were not known to have diabetes. The qualifying OGTT could be obtained up to 4 weeks prior to screening provided that anti-diabetic therapy (if any) remained unchanged between the qualifying OGTT and the screening visit. Two plasma glucose values were drawn during the OGTT - a fasting value (FPG) and a value drawn two hours after the 75 g oral glucose load was administered (postprandial plasma glucose [PPG]).

- Impaired glucose tolerance (IGT), defined as a PPG value ≥140 and <200 mg/dL (ie, ≥7.8 and <11.1 mmol/L), with a FPG <126 mg/dL (7.0 mmol/L).

OR

- Impaired fasting glucose (IFG), defined as an FPG ≥110 and <126 mg/dL (≥6.1 and <7 mmol/L), without diabetes mellitus (PPG must be <200 mg/dL [11.1 mmol/L]).

OR

- Early type 2 diabetes, defined as a FPG ≥126 mg/dL (7.0 mmol/L) or a PPG of ≥200 mg/dL (11.1 mmol/L), or a previous diagnosis of diabetes, and either:

* on no pharmacological treatment (while ambulatory) for at least 10 weeks prior to screening, with screening glycated hemoglobin <150% of the upper limit of normal (ULN) for the laboratory (eg, <9% if the ULN is 6%)
* or taking one oral antidiabetic drug (OAD) from among sulfonylureas (SU), biguanides, thiazolidinediones (TZDs), alpha-glucosidase inhibitors (AGIs), and meglitinides (MGTs) at a stable dose while ambulatory for at least 10 weeks at the time of screening (or for the 10 weeks prior to hospitalization if identified while hospitalized for a CV event), with screening glycated hemoglobin <133% of the ULN for the laboratory (eg, <8% if the ULN is 6%) if taking this medication at half-maximum dose or greater, and glycated hemoglobin <142% of the ULN for the laboratory (eg, <8.5% if the ULN is 6%) if taking this medication at less than half-maximum dose. Individuals taking combination products containing two or more OADs were not eligible.

I2. Men or women aged 50 years and older

I3. At least one of the following CV risk factors:

* previous myocardial infarction (MI) (≥ 5 days prior to randomization)
* previous stroke (≥ 5 days prior to randomization)
* previous coronary, carotid or peripheral arterial revascularization
* angina with documented ischemic changes (at least 2 mm ST segment depression on electrocardiogram during a Graded Exercise Test [GXT]; or with a cardiac imaging study positive for ischemia); or unstable angina with documented ischemic changes (either ST segment depression of at least 1 mm or an increase in troponin above the normal range but below the range diagnostic for acute myocardial infarction)
* microalbuminuria or clinical albuminuria (an albumin: creatinine ratio ≥ 30 μg/mg in at least one or timed collection of urine with albumin excretion ≥20 μg/min or ≥30 mg/24 hours or total protein excretion ≥500 mg/24 hours)
* left ventricular hypertrophy by electrocardiogram or echocardiogram
* significant stenosis on angiography of coronary, carotid, or lower extremity arteries (ie, 50% or more stenosis)
* ankle-brachial index < 0.9.

I4. Provision of signed and dated informed consent prior to any study procedures.

I5. Ability and willingness to complete study diaries and questionnaires.

I6. Demonstrated ability to use the self-glucose-monitoring device, and to self-inject insulin prior to randomization.

I7. A negative pregnancy test for all women of childbearing potential (ie, ovulating, pre- menopausal, and not surgically sterile) and the agreement of these women to use a reliable method of birth control to prevent pregnancy during the duration of the study .

I8. Willingness to discontinue prior omega-3 PUFA supplements for the duration of the study.

Exclusion criteria

E1. Type 1 diabetes.

E2. Requiring ambulatory insulin treatment or uncontrolled or symptomatic hyperglycemia that is likely to require the addition of ambulatory insulin therapy or a new antidiabetic agent either before or within 2 weeks after randomization.

E3. Known anti-glutamic acid decarboxylase antibody (anti-GAD Ab) positivity in the past.

E4. Screening glycated hemoglobin ≥150% of the ULN for the laboratory (eg, ≥9% if the ULN is 6%).

E5. Unwillingness to inject insulin or perform self-monitoring of blood glucose.

E6. Nonadherence to the run-in requirement to inject placebo insulin and do capillary glucose monitoring for at least 4 days prior to randomization.

E7. Coronary artery bypass grafting (CABG) either planned at the time of screening, or CABG within the 4 years prior to screening - however, participants with angina, MI, or stroke since a previous CABG will be eligible for randomization, even if the last CABG was within 4 years.

E8. Serum creatinine >2.0 mg/dL (176 μmol/L) at screening.

E9. Active liver disease, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 times ULN at screening.

E10. Chronic or recurrent treatment with systemic corticosteroids, or niacin treatment for hyperlipidemia.

E11. Heart failure of New York Heart Association (NYHA) Functional Class III or IV.

E12. Expected survival of <3 years for non-CV causes such as cancer.

E13. Any other factor likely to limit protocol compliance or reporting of adverse events (AEs).

E14. Unwilling or unable to discontinue TZDs.

E15. Simultaneous participation in any other clinical trial of an active pharmacologic agent.

E16. Unwillingness to permit sites to contact their primary physicians to communicate information about the study and the participant's data and treatment assignment.

E17. History of hypersensitivity to the investigational products.

E18. Previous randomization in this study.

E19. A prior heart transplant, or awaiting a heart transplant.

E20. Known infection with human immunodeficiency virus (HIV).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12537 (Actual)
Dates: Start 2003-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi; Hertzel Gerstein, M.D., Principal Investigator — McMaster University and Hamilton Health Sciences; Salim Yusuf, M.D., Principal Investigator — McMaster University and Hamilton Health Sciences
Locations (40):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Cove, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Minsk, Belarus
- Sanofi-Aventis Administrative Office, Hamilton, Bermuda
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Beijing, China
- Sanofi-Aventis Administrative Office, Cali, Colombia
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Tatari, Estonia
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Makati City, Dublin, Ireland
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Riga, Latvia
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Aministrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford, Surrey, United Kingdom
- Makati City, Caracas, Venezuela

REFERENCES:
- [Background] Origin Trial Investigators; Gerstein H, Yusuf S, Riddle MC, Ryden L, Bosch J. Rationale, design, and baseline characteristics for a large international trial of cardiovascular disease prevention in people with dysglycemia: the ORIGIN Trial (Outcome Reduction with an Initial Glargine Intervention). Am Heart J. 2008 Jan;155(1):26-32, 32.e1-6. doi: 10.1016/j.ahj.2007.09.009. Epub 2007 Nov 26. PMID 18082485
- [Background] Hanefeld M, Koehler C, Hoffmann C, Wilhelm K, Kamke W, Gerstein H. Effect of targeting normal fasting glucose levels with basal insulin glargine on glycaemic variability and risk of hypoglycaemia: a randomized, controlled study in patients with early Type 2 diabetes. Diabet Med. 2010 Feb;27(2):175-80. doi: 10.1111/j.1464-5491.2009.02915.x. PMID 20546261
- [Background] Badings EA, Dyal L, Schoterman L, Lok DJ, Stoel I, Gerding MN, Gerstein HC, Tijssen JG. Strategies to detect abnormal glucose metabolism in people at high risk of cardiovascular disease from the ORIGIN (Outcome Reduction with Initial Glargine Intervention) trial population. J Diabetes. 2011 Sep;3(3):232-7. doi: 10.1111/j.1753-0407.2011.00124.x. PMID 21631894
- [Background] Ramachandran A, Riddle MC, Kabali C, Gerstein HC; ORIGIN Investigators. Relationship between A1C and fasting plasma glucose in dysglycemia or type 2 diabetes: an analysis of baseline data from the ORIGIN trial. Diabetes Care. 2012 Apr;35(4):749-53. doi: 10.2337/dc11-1918. Epub 2012 Feb 8. PMID 22323416
- [Result] ORIGIN Trial Investigators; Gerstein HC, Bosch J, Dagenais GR, Diaz R, Jung H, Maggioni AP, Pogue J, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. Basal insulin and cardiovascular and other outcomes in dysglycemia. N Engl J Med. 2012 Jul 26;367(4):319-28. doi: 10.1056/NEJMoa1203858. Epub 2012 Jun 11. PMID 22686416
- [Result] ORIGIN Trial Investigators; Bosch J, Gerstein HC, Dagenais GR, Diaz R, Dyal L, Jung H, Maggiono AP, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. n-3 fatty acids and cardiovascular outcomes in patients with dysglycemia. N Engl J Med. 2012 Jul 26;367(4):309-18. doi: 10.1056/NEJMoa1203859. Epub 2012 Jun 11. PMID 22686415
- [Derived] Lee SF, Ramasundarahettige C, Gerstein HC, McIntyre WF, Eikelboom J, O'Donnell MJ, Zhou Y, Bangdiwala SI, Thabane L. Comparison of total event analysis and first event analysis in relation to heterogeneity in cardiovascular trials. BMC Med Res Methodol. 2025 Jun 9;25(1):159. doi: 10.1186/s12874-025-02593-3. PMID 40490702
- [Derived] Pigeyre M, Gerstein H, Ahlqvist E, Hess S, Pare G. Identifying blood biomarkers for type 2 diabetes subtyping: a report from the ORIGIN trial. Diabetologia. 2023 Jun;66(6):1045-1051. doi: 10.1007/s00125-023-05887-7. Epub 2023 Mar 1. PMID 36854916
- [Derived] Cukierman-Yaffe T, Lee SF, Pare G, McQueen M, Hess S, Gerstein HC. Biomarkers of Prevalent and Incident Cognitive Dysfunction in People with Dysglycemia: Data from the ORIGIN Trial. J Alzheimers Dis. 2022;87(3):1143-1150. doi: 10.3233/JAD-215195. PMID 35431237
- [Derived] Shao H, Kianmehr H, Guo J, Li P, Fonseca V, Shi L. Efficacy of iGlarLixi on 5-year risk of diabetes-related complications: A simulation study. J Diabetes Complications. 2022 Mar;36(3):108132. doi: 10.1016/j.jdiacomp.2022.108132. Epub 2022 Jan 25. PMID 35101326
- [Derived] Pigeyre M, Hess S, Gomez MF, Asplund O, Groop L, Pare G, Gerstein H. Validation of the classification for type 2 diabetes into five subgroups: a report from the ORIGIN trial. Diabetologia. 2022 Jan;65(1):206-215. doi: 10.1007/s00125-021-05567-4. Epub 2021 Oct 21. PMID 34676424
- [Derived] Wang A, Gerstein HC, Lee SF, Hess S, Pare G, Ryden L, Mellbin LG. Testosterone and sex hormone-binding globulin in dysglycemic women at high cardiovascular risk: A report from the Outcome Reduction with an Initial Glargine Intervention trial. Diab Vasc Dis Res. 2021 Mar-Apr;18(2):14791641211002475. doi: 10.1177/14791641211002475. PMID 33752449
- [Derived] Pigeyre M, Sjaarda J, Chong M, Hess S, Bosch J, Yusuf S, Gerstein H, Pare G. ACE and Type 2 Diabetes Risk: A Mendelian Randomization Study. Diabetes Care. 2020 Apr;43(4):835-842. doi: 10.2337/dc19-1973. Epub 2020 Feb 4. PMID 32019855
- [Derived] Theriault S, Sjaarda J, Chong M, Hess S, Gerstein H, Pare G. Identification of Circulating Proteins Associated With Blood Pressure Using Mendelian Randomization. Circ Genom Precis Med. 2020 Feb;13(1):e002605. doi: 10.1161/CIRCGEN.119.002605. Epub 2020 Jan 12. PMID 31928076
- [Derived] Gerstein HC, Pare G, McQueen MJ, Lee SF, Bangdiwala SI, Kannt A, Hess S; ORIGIN Trial Investigators. Novel Biomarkers for Change in Renal Function in People With Dysglycemia. Diabetes Care. 2020 Feb;43(2):433-439. doi: 10.2337/dc19-1604. Epub 2019 Nov 14. PMID 31727687
- [Derived] Pigeyre M, Sjaarda J, Mao S, Chong M, Hess S, Yusuf S, Gerstein H, Pare G. Identification of Novel Causal Blood Biomarkers Linking Metabolically Favorable Adiposity With Type 2 Diabetes Risk. Diabetes Care. 2019 Sep;42(9):1800-1808. doi: 10.2337/dc18-2444. Epub 2019 Jun 24. PMID 31235487
- [Derived] Cukierman-Yaffe T, Bosch J, Jung H, Punthakee Z, Gerstein HC. Hypoglycemia and Incident Cognitive Dysfunction: A Post Hoc Analysis From the ORIGIN Trial. Diabetes Care. 2019 Jan;42(1):142-147. doi: 10.2337/dc18-0690. Epub 2018 Nov 13. PMID 30425095
- [Derived] Mohammadi-Shemirani P, Sjaarda J, Gerstein HC, Treleaven DJ, Walsh M, Mann JF, McQueen MJ, Hess S, Pare G. A Mendelian Randomization-Based Approach to Identify Early and Sensitive Diagnostic Biomarkers of Disease. Clin Chem. 2019 Mar;65(3):427-436. doi: 10.1373/clinchem.2018.291104. Epub 2018 Oct 18. PMID 30337280
- [Derived] Morieri ML, Gao H, Pigeyre M, Shah HS, Sjaarda J, Mendonca C, Hastings T, Buranasupkajorn P, Motsinger-Reif AA, Rotroff DM, Sigal RJ, Marcovina SM, Kraft P, Buse JB, Wagner MJ, Gerstein HC, Mychaleckyj JC, Pare G, Doria A. Genetic Tools for Coronary Risk Assessment in Type 2 Diabetes: A Cohort Study From the ACCORD Clinical Trial. Diabetes Care. 2018 Nov;41(11):2404-2413. doi: 10.2337/dc18-0709. Epub 2018 Sep 27. PMID 30262460
- [Derived] Birkeland KI, Grill V, Wium C, McQueen MJ, Lopez-Jaramillo P, Lee SF, Gerstein HC. The association of basal insulin treatment versus standard care with outcomes in anti-GAD positive and negative subjects: A post-hoc analysis of the ORIGIN trial. Diabetes Obes Metab. 2019 Feb;21(2):429-433. doi: 10.1111/dom.13528. Epub 2018 Oct 3. PMID 30203580
- [Derived] Sjaarda J, Gerstein H, Chong M, Yusuf S, Meyre D, Anand SS, Hess S, Pare G. Blood CSF1 and CXCL12 as Causal Mediators of Coronary Artery Disease. J Am Coll Cardiol. 2018 Jul 17;72(3):300-310. doi: 10.1016/j.jacc.2018.04.067. Epub 2018 Jul 9. PMID 30012324
- [Derived] Gerstein HC, Ferrannini E, Riddle MC, Yusuf S; ORIGIN Trial Investigators. Insulin resistance and cardiovascular outcomes in the ORIGIN trial. Diabetes Obes Metab. 2018 Mar;20(3):564-570. doi: 10.1111/dom.13112. Epub 2017 Oct 8. PMID 28895655
- [Derived] Papademetriou V, Nylen ES, Doumas M, Probstfield J, Mann JFE, Gilbert RE, Gerstein HC. Chronic Kidney Disease, Basal Insulin Glargine, and Health Outcomes in People with Dysglycemia: The ORIGIN Study. Am J Med. 2017 Dec;130(12):1465.e27-1465.e39. doi: 10.1016/j.amjmed.2017.05.047. Epub 2017 Aug 31. PMID 28842165
- [Derived] Yates T, Davies MJ, Jung H, Bosch J, Spinas GA, Sreenan S, Commerford P, Gerstein HC; ORGIN investigators. Effect of insulin glargine on recreational physical activity and TV viewing: Analysis of the randomised ORIGIN trial. Diabetes Res Clin Pract. 2017 Oct;132:137-143. doi: 10.1016/j.diabres.2017.07.035. Epub 2017 Jul 31. PMID 28837885
- [Derived] Rautio A, Boman K, Gerstein HC, Hernestal-Boman J, Lee SF, Olofsson M, Mellbin LG. The effect of basal insulin glargine on the fibrinolytic system and von Willebrand factor in people with dysglycaemia and high risk for cardiovascular events: Swedish substudy of the Outcome Reduction with an Initial Glargine Intervention trial. Diab Vasc Dis Res. 2017 Jul;14(4):345-352. doi: 10.1177/1479164117703034. Epub 2017 Apr 12. PMID 28403644
- [Derived] Gerstein HC, Pare G, McQueen MJ, Lee SF, Hess S; ORIGIN Trial Investigators. Validation of the ORIGIN Cardiovascular Biomarker Panel and the Value of Adding Troponin I in Dysglycemic People. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2251-2257. doi: 10.1210/jc.2017-00273. PMID 28368516
- [Derived] Gerstein HC, Pare G, Hess S, Ford RJ, Sjaarda J, Raman K, McQueen M, Lee S, Haenel H, Steinberg GR; ORIGIN Investigators. Growth Differentiation Factor 15 as a Novel Biomarker for Metformin. Diabetes Care. 2017 Feb;40(2):280-283. doi: 10.2337/dc16-1682. Epub 2016 Dec 14. PMID 27974345
- [Derived] ORIGIN Trial Investigators. Cardiovascular and Other Outcomes Postintervention With Insulin Glargine and Omega-3 Fatty Acids (ORIGINALE). Diabetes Care. 2016 May;39(5):709-16. doi: 10.2337/dc15-1676. Epub 2015 Dec 17. PMID 26681720
- [Derived] Gerstein HC, Pare G, McQueen MJ, Haenel H, Lee SF, Pogue J, Maggioni AP, Yusuf S, Hess S; Outcome Reduction With Initial Glargine Intervention Trial Investigators. Identifying Novel Biomarkers for Cardiovascular Events or Death in People With Dysglycemia. Circulation. 2015 Dec 15;132(24):2297-304. doi: 10.1161/CIRCULATIONAHA.115.015744. Epub 2015 Oct 30. PMID 26518765
- [Derived] Cukierman-Yaffe T, Bosch J, Diaz R, Dyal L, Hancu N, Hildebrandt P, Lanas F, Lewis BS, Marre M, Yale JF, Yusuf S, Gerstein HC; ORIGIN Investigators. Effects of basal insulin glargine and omega-3 fatty acid on cognitive decline and probable cognitive impairment in people with dysglycaemia: a substudy of the ORIGIN trial. Lancet Diabetes Endocrinol. 2014 Jul;2(7):562-72. doi: 10.1016/S2213-8587(14)70062-2. Epub 2014 Jun 2. PMID 24898834
- [Derived] ORIGIN trial investigators; Gilbert RE, Mann JF, Hanefeld M, Spinas G, Bosch J, Yusuf S, Gerstein HC. Basal insulin glargine and microvascular outcomes in dysglycaemic individuals: results of the Outcome Reduction with an Initial Glargine Intervention (ORIGIN) trial. Diabetologia. 2014 Jul;57(7):1325-31. doi: 10.1007/s00125-014-3238-4. Epub 2014 Apr 26. PMID 24771090
- [Derived] Lopez-Jaramillo P, Cohen DD, Gomez-Arbelaez D, Bosch J, Dyal L, Yusuf S, Gerstein HC; ORIGIN Trial Investigators. Association of handgrip strength to cardiovascular mortality in pre-diabetic and diabetic patients: a subanalysis of the ORIGIN trial. Int J Cardiol. 2014 Jun 15;174(2):458-61. doi: 10.1016/j.ijcard.2014.04.013. Epub 2014 Apr 13. No abstract available. PMID 24768457
- [Derived] Lamy A, Tong W, Jung H, Gafni A, Singh K, Tyrwhitt J, Yusuf S, Gerstein HC; ORIGIN Investigators. Cost implications of the use of basal insulin glargine in people with early dysglycemia: the ORIGIN trial. J Diabetes Complications. 2014 Jul-Aug;28(4):553-8. doi: 10.1016/j.jdiacomp.2014.02.012. Epub 2014 Mar 2. PMID 24684774
- [Derived] Bordeleau L, Yakubovich N, Dagenais GR, Rosenstock J, Probstfield J, Chang Yu P, Ryden LE, Pirags V, Spinas GA, Birkeland KI, Ratner RE, Marin-Neto JA, Keltai M, Riddle MC, Bosch J, Yusuf S, Gerstein HC; ORIGIN Trial Investigators. The association of basal insulin glargine and/or n-3 fatty acids with incident cancers in patients with dysglycemia. Diabetes Care. 2014;37(5):1360-6. doi: 10.2337/dc13-1468. Epub 2014 Feb 26. PMID 24574355
- [Derived] ORIGIN Trial Investigators; Mellbin LG, Ryden L, Riddle MC, Probstfield J, Rosenstock J, Diaz R, Yusuf S, Gerstein HC. Does hypoglycaemia increase the risk of cardiovascular events? A report from the ORIGIN trial. Eur Heart J. 2013 Oct;34(40):3137-44. doi: 10.1093/eurheartj/eht332. Epub 2013 Sep 2. PMID 23999452
- [Derived] ORIGIN Trial Investigators. Characteristics associated with maintenance of mean A1C<6.5% in people with dysglycemia in the ORIGIN trial. Diabetes Care. 2013 Oct;36(10):2915-22. doi: 10.2337/dc12-2238. Epub 2013 May 8. PMID 23656980
- [Derived] Lonn EM, Bosch J, Diaz R, Lopez-Jaramillo P, Ramachandran A, Hancu N, Hanefeld M, Krum H, Ryden L, Smith S, McQueen MJ, Dyal L, Yusuf S, Gerstein HC; GRACE and ORIGIN Investigators. Effect of insulin glargine and n-3FA on carotid intima-media thickness in people with dysglycemia at high risk for cardiovascular events: the glucose reduction and atherosclerosis continuing evaluation study (ORIGIN-GRACE). Diabetes Care. 2013 Sep;36(9):2466-74. doi: 10.2337/dc12-2129. Epub 2013 Apr 5. PMID 23564916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 575 sites in 40 countries between August 22, 2003 and December 19, 2011. Three sites were closed and data from these sites were not analyzed following site audits and in compliance with rulings from national health authorities.
Pre-assignment Details: The purpose of the factorial design was to efficiently answer two independent scientifically worthwhile questions regarding insulin glargine and omega-3 fatty acids within the context of a single clinical trial. Sample size was determined based on the insulin glargine study objective. Results reported below are those of the insulin glargine study.
Groups:
- Insulin Glargine: Treatment with Insulin Glargine with or without omega-3 polyunsaturated fatty acids
- Standard Care: Standard care with or without omega-3 polyunsaturated fatty acids
Period: Overall Study
Arm/Group | Insulin Glargine | Standard Care
Started | 6264 (randomized participants = intent-to-treat (ITT) population) | 6273 (randomized participants = intent-to-treat (ITT) population)
Safety Population (Treated) | 6231 (randomized patients who received at least one dose of insulin glargine) | 6273 (patients randomized to standard care arm)
Completed | 5052 (completed study treatment) | 6273 (not applicable (no treatment))
Not Completed | 1212 | 0
Not completed — Adverse Event | 105 | 0
Not completed — Withdrawal by Subject | 1090 | 0
Not completed — Other | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine | Standard Care | Total
Number analyzed (Participants) | 6264 | 6273 | 12537
Age Continuous [Mean (Standard Deviation); unit: years] | 63.5 (7.8) | 63.5 (7.9) | 63.5 (7.8)
Sex/Gender, Customized [Number; unit: participants]
  Male | 4181 | 3969 | 8150
  Female | 2082 | 2304 | 4386
  Missing value | 1 | 0 | 1
Baseline Weight [Mean (Standard Deviation); unit: kg] — Due to missing values, N=6256 for insulin glargine and N=6271 for standard care.
  kg | 83.33 (16.77) | 83.13 (17.28) | 83.23 (17.03)
Baseline Body Mass Index [Mean (Standard Deviation); unit: kg/m²] — Due to missing values, N=6251 for insulin glargine and N=6270 for standard care.
  kg/m² | 29.77 (5.17) | 29.88 (5.33) | 29.82 (5.25)
Any previous cardiovascular event [Number; unit: participants]
  No | 2552 | 2607 | 5159
  Yes | 3712 | 3666 | 7378
Diabetes diagnosis at time of screening [Number; unit: participants] — IFG = Impaired Fasting Glucose defined as a Postprandial Plasma Glucose (PPG) value ≥140 and <200 mg/dL (ie, ≥7.8 and <11.1 mmol/L), with a Fasting Plasma Glucose (FPG) <126 mg/dL (7.0 mmol/L)
  IGT = Impaired Glucose Tolerance defined as an FPG ≥110 and <126 mg/dL (≥6.1 and <7 mmol/L), without diabetes mellitus (PPG must be <200 mg/dL [11.1 mmol/L])
  OAD = oral antidiabetic drug
  participants
    IFG and/or IGT | 735 | 717 | 1452
    Newly diagnosed diabetic | 365 | 395 | 760
    Established diabetes with no OAD treatment | 1414 | 1467 | 2881
    Established diabetes with one OAD treatment | 3748 | 3692 | 7440
    Unclear diabetes status | 2 | 2 | 4
Duration of diabetes for established diabetes patients [Median (Inter-Quartile Range); unit: years] — Population of patients with established diabetes. Due to missing values, N=5148 for insulin glargine and N=5141 for standard care.
  years | 3.50 [1.50 to 7.50] | 3.50 [1.50 to 7.50] | 3.50 [1.50 to 7.50]
Glycated Hemoglobin A1c (HbA1c) [Median (Inter-Quartile Range); unit: percent] — Due to missing values, N=6175 for insulin glargine and N=6189 for standard care.
  percent | 6.41 [5.81 to 7.18] | 6.40 [5.81 to 7.16] | 6.40 [5.81 to 7.18]
Fasting Plasma Glucose [Median (Inter-Quartile Range); unit: mmol/L] — Due to missing values, N=6248 for insulin glargine and N=6266 for standard care.
  mmol/L | 6.94 [6.05 to 8.20] | 6.90 [6.00 to 8.20] | 6.94 [6.05 to 8.20]

OUTCOME MEASURES:

1. Primary Outcome: Composite of the First Occurrence of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI) or Nonfatal Stroke
Description: Number of participants with a first occurrence of one of the above events.
  The outcome's evaluation is based on the number of such positively-adjudicated first events occurring for patients assigned to the study groups. Assessments of the above events were reviewed by the Event Adjudication Committee who was kept blinded to the group assignment of participants.
  Statistical analysis is performed on the time from randomization to the first occurrence of the events. Number of participants with a composite endpoint (i.e. with first occurrence of CV death, nonfatal MI or nonfatal stroke) is provided in the first row of the statistical table.
Time Frame: from randomization until study cut-off date (median duration of follow-up: 6.2 years)
Population: The analysis was based on the intent-to-treat (ITT) population i.e. all randomized participants.
  For the endpoint's composition, the numbers only summarize the event when it was the first occurrence of the endpoint. A participant is counted only once within a category. The same participant may appear in different categories.
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Standard Care
Number analyzed (Participants) | 6264 | 6273
participants
  Participants with a composite endpoint | 1041 | 1013
  Endpoint's composition: CV death | 484 | 476
  Endpoint's composition: nonfatal MI | 297 | 282
  Endpoint's composition: nonfatal stroke | 261 | 256
Statistical Analysis 1: Comparison: Insulin Glargine vs Standard Care; The total required number of first coprimary outcomes (2200) assumed that a hazard reduction of 14-16% was clinically significant and controlled the overall experiment-wise Type 1 error at 5% with a power of 80% for each outcome. The total number of participants needed to achieve this number of events within the planned enrollment and treatment periods was ultimately estimated to be 12 500 based on the CURE and HOPE study databases; Test type: Superiority or Other; p = 0.6273, Log Rank — For the analysis of the two coprimary efficacy outcomes, the overall Type 1 error was partitioned. The first coprimary outcome was tested at 4.4%, whereas the second coprimary outcome was tested at 1% (weighted Hochberg procedure); Log-rank test stratified by double-blind treatment (omega-3 PUFA, placebo), baseline diabetes diagnosis and previous CV event; Cox Proportional Hazard = 1.022, 95% CI 2-sided [0.937 to 1.114] — Hazard ratio (glargine/standard care) estimated by Cox regression model with treatment (glargine, standard care) as factor, stratified by double-blind treatment (omega-3 PUFA, placebo), baseline diabetes diagnosis and previous CV event

2. Primary Outcome: Composite of the First Occurrence of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), Nonfatal Stroke, Revascularization Procedure or Hospitalization for Heart Failure (HF)
Description: Number of participants with a first occurrence of one of the above events (revascularization procedures included coronary artery bypass graft, percutaneous transluminal coronary angioplasty (PTCA) i.e. balloon, PTCA with stent, other percutaneous intervention, carotid angioplasty with/without stent, carotid endarterectomy, peripheral angioplasty with or without stent, peripheral vascular surgery, and limb amputation due to vascular disease).
  The outcome's evaluation is based on the number of such positively-adjudicated first events occurring for patients assigned to the study groups. Assessments of the above events were reviewed by the Event Adjudication Committee who was kept blinded to the group assignment of participants.
  Statistical analysis is performed on the time from randomization to the first occurrence of the events. Number of participants with a composite endpoint (i.e. with first occurrence of the events) is provided in the first row of the statistical table.
Time Frame: from randomization until study cut-off date (median duration of follow-up: 6.2 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Standard Care
Number analyzed (Participants) | 6264 | 6273
participants
  Participants with a composite endpoint | 1792 | 1727
  Endpoint's composition: CV death | 350 | 339
  Endpoint's composition: nonfatal MI | 257 | 238
  Endpoint's composition: nonfatal stroke | 231 | 227
  Endpoint's composition: revascularization | 763 | 717
  Endpoint's composition: hospitalization for HF | 249 | 259
Statistical Analysis 1: Comparison: Insulin Glargine vs Standard Care; See above additional details provided for the analysis of the first coprimary outcome; Test type: Superiority or Other; p = 0.2692, Log Rank — The second coprimary outcome was tested at 1% (see above additional information for the first coprimary outcome); [statistical method as in outcome 1, analysis 1]; Cox Proportional Hazard = 1.038, 95% CI 2-sided [0.972 to 1.109] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Total Mortality (All Causes)
Description: Number of deaths due to any cause
Time Frame: from randomization until study cut-off date (median duration of follow-up: 6.2 years)
Population: The analysis was based on the intent-to-treat (ITT) population, which was all randomized participants, regardless of compliance with the protocol.
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Standard Care
Number analyzed (Participants) | 6264 | 6273
participants | 951 | 965
Statistical Analysis 1: Comparison: Insulin Glargine vs Standard Care; Test type: Superiority or Other; Cox Proportional Hazard = 0.983, 95% CI 2-sided [0.899 to 1.076] — Hazard ratio (glargine/standard care) estimated by Cox regression model with treatment (glargine, standard care) as factor, with double-blind treatment (omega-3 PUFA, placebo), baseline diabetes diagnosis and previous CV event as covariates

4. Secondary Outcome: Composite Diabetic Microvascular Outcome (Kidney or Eye Disease)
Description: The composite outcome used to analyze microvascular disease progression contained components of clinical events:
  * the occurrence of laser surgery or vitrectomy for diabetic retinopathy (DR);
  * the development of blindness due to DR;
  * the occurrence of renal death or renal replacement therapy; as well as the following laboratory-based events:
  * doubling of serum creatinine; or
  * progression of albuminuria (from none to microalbuminuria [at least 30 mg/g creatinine], to macroalbuminuria [at least 300 mg/g creatinine]).
Time Frame: from randomization until study cut-off date (median duration of follow-up: 6.2 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Standard Care
Number analyzed (Participants) | 6264 | 6273
participants
  Participants with a composite endpoint | 1323 | 1363
  Endpoint's composition: vitrectomy | 24 | 25
  Endpoint's composition: laser therapy for DR | 57 | 67
  Endpoint's composition: dialysis | 18 | 28
  Endpoint's composition: renal transplant | 0 | 0
  Endpoint's composition: serum creatinine doubled | 82 | 88
  Endpoint's composition: death due to renal failure | 4 | 3
  Endpoint's composition: albuminuria progression | 1153 | 1171
Statistical Analysis 1: Comparison: Insulin Glargine vs Standard Care; Test type: Superiority or Other; Cox Proportional Hazard = 0.970, 95% CI 2-sided [0.900 to 1.047] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Incidence of Development of Type 2 Diabetes Mellitus in Participants With IGT and/or IFG
Description: The incidence was determined by calculating the proportion of randomized participants without diabetes at randomization who either developed diabetes during the study or who were classified as having possible diabetes based on results of two oral glucose tolerance tests (OGTT) performed after the last follow-up visit (within 21-28 days for OGTT#1 and within 10-14 weeks for OGTT#2).
Time Frame: from randomization until the last follow-up visit or last OGTT (median duration of follow-up: 6.2 years)
Population: The analysis was based on the subgroup of the intent-to-treat (ITT) population without diabetes at randomization.
Measure: Number; unit: percentage of patients
Arm/Group | Insulin Glargine | Standard Care
Number analyzed (Participants) | 737 | 719
percentage of patients | 24.7 | 31.2
Statistical Analysis 1: Comparison: Insulin Glargine vs Standard Care; Test type: Superiority or Other; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.58 to 0.91] — Odds ratio estimated using Cochran-Mantel-Haenszel (CMH) test method stratified by double-blind treatment (omega-3 PUFA or placebo) and previous cardiovascular event (yes or no)

6. Other Pre Specified Outcome: Number of Patients With Various Types of Symptomatic Hypoglycemia Events
Description: Symptomatic hypoglycemia was defined as an event with clinical symptoms consistent with hypoglycemia, based on data recorded in the participant's diary. These were further categorized as confirmed (ie, with a concomitant home glucose reading ≤54 mg/dL [≤3.0 mmol/L]) or unconfirmed.
  Severe hypoglycemia was defined as an event with clinical symptoms consistent with hypoglycemia in which the participant required the assistance of another person, and one of the following:
  * the event was associated with a documented self-measured or laboratory plasma glucose level ≤36 mg/dL (≤2.0 mmol/L), or
  * the event was associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration.
Time Frame: on-treatment period (median duration of follow-up: 6.2 years)
Population: The population analyzed was the safety population consisting of all randomized and treated patients (who received at least one dose of study drug) for the insulin glargine group and of all randomized patients for the standard care group.
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Standard Care
Number analyzed (Participants) | 6231 | 6273
participants
  Patients with hypoglycemia events | 3597 | 1624
  Patients with non-severe hypoglycemia | 3533 | 1582
  Patients with confirmed non-severe hypoglycemia | 2581 | 904
  Patients with severe hypoglycemia | 352 | 113

7. Other Pre Specified Outcome: Number of Patients With First Occurrence of Any Type of Cancer
Description: Data on cancers that occurred in association with hospitalizations were collected systematically in both groups from the start of the study. All reported cancers occurring during the trial (new or recurrent) were adjudicated by the Event Adjudication Committee.
Time Frame: from randomization until study cut-off date (median duration of follow-up: 6.2 years)
Population: The analysis was based on the intent-to-treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Insulin Glargine | Standard Care
Number analyzed (Participants) | 6264 | 6273
participants | 559 | 561

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed through the study. The median duration of follow-up was 6.2 years.
Description: Aside from hypoglycemia and cancer, serious AEs were only captured if the event was considered related to a study drug. Non-serious AEs were only captured if the event resulted in some modification (suspension, alteration or cessation) in the dose of a study drug. This creates a bias for the comparison between insulin glargine and standard care.
Arm/Group | Insulin Glargine | Standard Care
Serious Adverse Events (participants affected / at risk) | 303/6231 | 232/6273
Other Adverse Events (participants affected / at risk) | 0/6231 | 0/6273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine (N=6231) | Standard Care (N=6273)
Pneumonia (Infections and infestations) | 5 | 6
Gastroenteritis (Infections and infestations) | 2 | 3
Sepsis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 4
Cellulitis (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic neoplasm malignant non-resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pseudomyxoma peritonei (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 36 | 15
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 21 | 0
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 7 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Hypomania (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 18 | 2
Cerebrovascular accident (Nervous system disorders) | 8 | 5
Syncope (Nervous system disorders) | 4 | 1
Cerebral haemorrhage (Nervous system disorders) | 3 | 0
Grand mal convulsion (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cranial nerve palsies multiple (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Vitreous haemorrhage (Eye disorders) | 2 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Retinal oedema (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Eversion of lacrimal punctum (Eye disorders) | 0 | 1
Retinal vein thrombosis (Eye disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 1
Otosclerosis (Ear and labyrinth disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 10 | 9
Angina unstable (Cardiac disorders) | 9 | 11
Acute myocardial infarction (Cardiac disorders) | 8 | 4
Cardiac failure congestive (Cardiac disorders) | 6 | 6
Arrhythmia supraventricular (Cardiac disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 3
Angina pectoris (Cardiac disorders) | 2 | 3
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 3
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial disease (Cardiac disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 3
Hypertensive emergency (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 1
Ischaemia (Vascular disorders) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal varices (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 2 | 1
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2
Nephropathy (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0
Skull malformation (Congenital, familial and genetic disorders) | 0 | 1
Death (General disorders) | 11 | 14
Chest pain (General disorders) | 6 | 2
Non-cardiac chest pain (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 3 | 0
Sudden death (General disorders) | 3 | 1
Cardiac death (General disorders) | 1 | 1
Device failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 1
Hernia obstructive (General disorders) | 0 | 1
Arteriogram coronary (Investigations) | 4 | 1
Weight increased (Investigations) | 2 | 0
Arteriogram carotid (Investigations) | 1 | 0
Biopsy lymph gland (Investigations) | 1 | 0
Colonoscopy (Investigations) | 1 | 0
Diagnostic procedure (Investigations) | 1 | 0
Ureteroscopy (Investigations) | 1 | 0
Cystoscopy (Investigations) | 0 | 1
Investigation (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 5 | 0
Fracture (Injury, poisoning and procedural complications) | 3 | 3
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 2 | 1
Coronary artery bypass (Surgical and medical procedures) | 2 | 1
Cholecystostomy (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Intestinal resection (Surgical and medical procedures) | 1 | 0
Urethral dilation procedure (Surgical and medical procedures) | 1 | 0
Vitrectomy (Surgical and medical procedures) | 1 | 0
Abdominal hernia repair (Surgical and medical procedures) | 0 | 1
Angioplasty (Surgical and medical procedures) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Colporrhaphy (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Parotidectomy (Surgical and medical procedures) | 0 | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"The Steering Committee will be responsible for preparing summaries of the study results for publication in the medical literature, and will have the right to submit such summaries for publication after a review by the sponsor. In such cases comments from the sponsor to the Steering Committee are to be provided within 15 working days. All comments will be carefully considered by the Steering Committee who nevertheless have the final decision on the content of the manuscript."